CLINICAL TRIAL: NCT01743677
Title: A PHASE 1, RANDOMIZED, PLACEBO- AND POSITIVE-CONTROLLED CROSS-OVER STUDY TO DETERMINE THE EFFECT OF SINGLE-DOSE CP-690,550 ON QTC INTERVAL IN HEALTHY VOLUNTEERS
Brief Title: CP-690,550 Thorough QTc Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: A3921028; 2007-004492-19 (EudraCT Number)
Record Dates: First submitted 2012-10-25; First posted 2012-12-06 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: TQT study; CP-690; 550
MeSH Terms: interventions — tofacitinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CP-690,550 100 mg (Experimental)
  Interventions: Drug: CP-690,550
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Moxifloxacin hydrochloride (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: CP-690,550 — Single dose 100 mg (5 x 20 mg tablets)
  Arms: CP-690,550 100 mg
Drug: Placebo — Single dose placebo tablets (5 tablets)
  Arms: Placebo
Drug: Moxifloxacin — Single dose Avelox 400 mg tablet
  Arms: Moxifloxacin hydrochloride

SUMMARY:
ICH E14 recommends that a thorough QT/QTc (TQT) study should be performed to determine whether intensive monitoring of QT interval in target patient populations is required during later stages of development. The current study is designed to ascertain whether CP-690,550 is associated with QTc prolongation.

DETAILED DESCRIPTION:
The current study is designed to ascertain whether CP-690,550 is associated with QTc prolongation

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Use of tobacco- or nicotine-containing products in excess of equivalent of 5 cigarettes per day.
* 12-lead ECG demonstrating QTc >450 msec or other clinically significant abnormalities at Screening.
* History of risk factors for QT prolongation or torsades de pointes.
* Pregnant or nursing women; women of childbearing potential unwilling or unable to use an acceptable method of nonhormonal contraception from at least 14 days prior to first dose until completion of follow-up.
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to first dose of trial medication.
* Any clinically significant infections within past 3 months or evidence of infection in past 7 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10-26 (Actual); Primary Completion 2008-02-07 (Actual); Study Completion 2008-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Clinical Research Unit, Brussels, Belgium
- Pfizer Clinical Research Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921028&StudyName=CP-690%2C550%20Thorough%20QTc%20Study%20

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 100 mg Then Placebo Then Moxifloxacin 400 mg: Single oral dose of CP-690,550 100 milligram (mg) (5 x 20 mg tablets) in first intervention period; followed by single oral dose of placebo matched to CP-690,550 tablets in second intervention period; and single oral dose of moxifloxacin 400 mg tablet in third intervention period. A washout period of at least 7 days was maintained between each intervention period.
- CP-690,550 100 mg Then Moxifloxacin 400 mg Then Placebo: Single oral dose of CP-690,550 100 mg (5 x 20 mg tablets) in first intervention period; followed by single oral dose of moxifloxacin 400 mg tablet in second intervention period; and single oral dose of placebo matched to CP-690,550 tablets in third intervention period. A washout period of at least 7 days was maintained between each intervention period.
- Placebo Then CP-690,550 100 mg Then Moxifloxacin 400 mg: Single oral dose of placebo matched to CP-690,550 tablets in first intervention period; followed by single oral dose of CP-690,550 100 mg (5 x 20 mg tablets) in second intervention period; and single oral dose of moxifloxacin 400 mg tablet in third intervention period. A washout period of at least 7 days was maintained between each intervention period.
- Placebo Then Moxifloxacin 400 mg Then CP-690,550 100 mg: Single oral dose of placebo matched to CP-690,550 tablets in first intervention period; followed by single oral dose of moxifloxacin 400 mg tablet in second intervention period; and single oral dose of CP-690,550 100 mg (5 x 20 mg tablets) in third intervention period. A washout period of at least 7 days was maintained between each intervention period.
- Moxifloxacin 400 mg Then CP-690,550 100 mg Then Placebo: Single oral dose of moxifloxacin 400 mg tablet in first intervention period; followed by single oral dose of CP-690,550 100 mg (5 x 20 mg tablets) in second intervention period; and single oral dose of placebo matched to CP-690,550 tablets in third intervention period. A washout period of at least 7 days was maintained between each intervention period.
- Moxifloxacin 400 mg Then Placebo Then CP-690,550 100 mg: Single oral dose of moxifloxacin 400 mg tablet in first intervention period; followed by single oral dose of placebo matched to CP-690,550 tablets in second intervention period; and single oral dose of CP-690,550 100 mg (5 x 20 mg tablets) in third intervention period. A washout period of at least 7 days was maintained between each intervention period.
Period: First Intervention Period
Arm/Group | CP-690,550 100 mg Then Placebo Then Moxifloxacin 400 mg | CP-690,550 100 mg Then Moxifloxacin 400 mg Then Placebo | Placebo Then CP-690,550 100 mg Then Moxifloxacin 400 mg | Placebo Then Moxifloxacin 400 mg Then CP-690,550 100 mg | Moxifloxacin 400 mg Then CP-690,550 100 mg Then Placebo | Moxifloxacin 400 mg Then Placebo Then CP-690,550 100 mg
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (at Least 7 Days)
Arm/Group | CP-690,550 100 mg Then Placebo Then Moxifloxacin 400 mg | CP-690,550 100 mg Then Moxifloxacin 400 mg Then Placebo | Placebo Then CP-690,550 100 mg Then Moxifloxacin 400 mg | Placebo Then Moxifloxacin 400 mg Then CP-690,550 100 mg | Moxifloxacin 400 mg Then CP-690,550 100 mg Then Placebo | Moxifloxacin 400 mg Then Placebo Then CP-690,550 100 mg
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | CP-690,550 100 mg Then Placebo Then Moxifloxacin 400 mg | CP-690,550 100 mg Then Moxifloxacin 400 mg Then Placebo | Placebo Then CP-690,550 100 mg Then Moxifloxacin 400 mg | Placebo Then Moxifloxacin 400 mg Then CP-690,550 100 mg | Moxifloxacin 400 mg Then CP-690,550 100 mg Then Placebo | Moxifloxacin 400 mg Then Placebo Then CP-690,550 100 mg
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (at Least 7 Days)
Arm/Group | CP-690,550 100 mg Then Placebo Then Moxifloxacin 400 mg | CP-690,550 100 mg Then Moxifloxacin 400 mg Then Placebo | Placebo Then CP-690,550 100 mg Then Moxifloxacin 400 mg | Placebo Then Moxifloxacin 400 mg Then CP-690,550 100 mg | Moxifloxacin 400 mg Then CP-690,550 100 mg Then Placebo | Moxifloxacin 400 mg Then Placebo Then CP-690,550 100 mg
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | CP-690,550 100 mg Then Placebo Then Moxifloxacin 400 mg | CP-690,550 100 mg Then Moxifloxacin 400 mg Then Placebo | Placebo Then CP-690,550 100 mg Then Moxifloxacin 400 mg | Placebo Then Moxifloxacin 400 mg Then CP-690,550 100 mg | Moxifloxacin 400 mg Then CP-690,550 100 mg Then Placebo | Moxifloxacin 400 mg Then Placebo Then CP-690,550 100 mg
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive any treatment (CP-690,550 100 mg first, moxifloxacin 400 mg first, or placebo first).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 0.25 Hour Post-Dose
Description: Triplicate 12-lead electrocardiogram (ECG) measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to the beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using the QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR). Data is reported as Least Squares (LS) mean difference (CP-690,550 minus Placebo, baseline-adjusted).
Time Frame: 0.25 hour post-dose
Population: ECG analysis set included all randomized and treated participants who had at least 1 post-dose ECG measurement in at least 1 period of the crossover.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Groups:
- CP-690,550 100 mg: Single oral dose of CP-690,550 100 mg (5 x 20 mg tablets) in any intervention period.
- Placebo: Single oral dose of placebo matched to CP-690,550 tablets in any intervention period.
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
milliseconds (msec) | 416.48 (0.8823) | 417.77 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = -1.29, 90% CI 2-sided [-3.15 to 0.56]

2. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 0.5 Hour Post-Dose
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The QT interval was adjusted for RR interval using the QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR). Data is reported as LS mean difference (CP-690,550 minus Placebo, baseline-adjusted).
Time Frame: 0.5 hour post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 414.70 (0.8823) | 416.12 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = -1.42, 90% CI 2-sided [-3.28 to 0.43]

3. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 1 Hour Post-Dose
Description: as for outcome 2
Time Frame: 1 hour post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 414.69 (0.8823) | 416.98 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = -2.29, 90% CI 2-sided [-4.15 to -0.44]

4. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 2 Hours Post-Dose
Description: as for outcome 2
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 413.70 (0.8823) | 415.05 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = -1.35, 90% CI 2-sided [-3.21 to 0.50]

5. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 4 Hours Post-Dose
Description: as for outcome 2
Time Frame: 4 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 416.83 (0.8823) | 415.76 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = 1.08, 90% CI 2-sided [-0.78 to 2.93]

6. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 8 Hours Post-Dose
Description: as for outcome 2
Time Frame: 8 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 409.25 (0.8823) | 408.39 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = 0.86, 90% CI 2-sided [-1.00 to 2.71]

7. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 12 Hours Post-Dose
Description: as for outcome 2
Time Frame: 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 411.39 (0.8823) | 410.24 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = 1.15, 90% CI 2-sided [-0.71 to 3.00]

8. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 16 Hours Post-Dose
Description: as for outcome 2
Time Frame: 16 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 415.87 (0.8823) | 413.72 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = 2.15, 90% CI 2-sided [0.29 to 4.00]

9. Primary Outcome: Mean Time-Matched Difference in QTcF Intervals Between CP-690,550 Compared to Placebo at 24 Hours Post-Dose
Description: as for outcome 2
Time Frame: 24 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 412.53 (0.8823) | 411.18 (0.8823)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = 1.35, 90% CI 2-sided [-0.50 to 3.21]

10. Secondary Outcome: Mean Time-Matched Difference in QTcF Intervals Between Moxifloxacin Compared to Placebo
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The QT interval was adjusted for RR interval using the QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR). Data is reported as LS mean difference (moxifloxacin minus Placebo, baseline-adjusted).
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- Moxifloxacin 400 mg: Single oral dose of moxifloxacin 400 mg tablet in any intervention period.
- Placebo: Single oral dose of placebo matched to moxifloxacin 400 mg in any intervention period.
Arm/Group | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec | 426.34 (0.8823) | 415.05 (0.8823)
Statistical Analysis 1: Comparison: Moxifloxacin 400 mg vs Placebo; Test type: Superiority; Least Squares Mean Difference = 11.29, 90% CI 2-sided [9.62 to 12.96]

11. Secondary Outcome: Mean Time-Matched Difference in QTcB Intervals Between CP-690,550 Compared to Placebo
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The QT interval was adjusted for RR interval using the QT and RR from each ECG by Bazett's formula (QTcB = QT divided by square root of RR). Data is reported as LS mean difference (CP-690,550 minus Placebo, baseline-adjusted).
Time Frame: 0.25, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | CP-690,550 100 mg | Placebo
Number analyzed (Participants) | 60 | 60
msec
  0.25 Hour Post-Dose | 416.40 (1.1139) | 416.24 (1.1139)
  0.5 Hour Post-Dose | 416.69 (1.1139) | 414.91 (1.1139)
  1 Hour Post-Dose | 417.98 (1.1139) | 414.99 (1.1139)
  2 Hours Post-Dose | 414.54 (1.1139) | 413.46 (1.1139)
  4 Hours Post-Dose | 417.26 (1.1139) | 415.10 (1.1139)
  8 Hours Post-Dose | 412.91 (1.1139) | 412.86 (1.1139)
  12 Hours Post-Dose | 416.76 (1.1139) | 416.27 (1.1139)
  16 Hours Post-Dose | 416.44 (1.1139) | 414.33 (1.1139)
  24 Hours Post-Dose | 413.93 (1.1139) | 413.14 (1.1139)
Statistical Analysis 1: Comparison: CP-690,550 100 mg vs Placebo; 0.25 hour post-dose; Test type: Superiority; Least Squares Mean Difference = 0.16, 90% CI 2-sided [-2.11 to 2.44]
Statistical Analysis 2: Comparison: CP-690,550 100 mg vs Placebo; 0.5 hour post-dose; Test type: Superiority; Least Squares Mean Difference = 1.78, 90% CI 2-sided [-0.49 to 4.06]
Statistical Analysis 3: Comparison: CP-690,550 100 mg vs Placebo; 1 hour post-dose; Test type: Superiority; Least Squares Mean Difference = 2.99, 90% CI 2-sided [0.71 to 5.26]
Statistical Analysis 4: Comparison: CP-690,550 100 mg vs Placebo; 2 hours post-dose; Test type: Superiority; Least Squares Mean Difference = 1.08, 90% CI 2-sided [-1.19 to 3.36]
Statistical Analysis 5: Comparison: CP-690,550 100 mg vs Placebo; 4 hours post-dose; Test type: Superiority; Least Squares Mean Difference = 2.16, 90% CI 2-sided [-0.11 to 4.44]
Statistical Analysis 6: Comparison: CP-690,550 100 mg vs Placebo; 8 hours post-dose; Test type: Superiority; Least Squares Mean Difference = 0.05, 90% CI 2-sided [-2.22 to 2.33]
Statistical Analysis 7: Comparison: CP-690,550 100 mg vs Placebo; 12 hours post-dose; Test type: Superiority; Least Squares Mean Difference = 0.49, 90% CI 2-sided [-1.79 to 2.76]
Statistical Analysis 8: Comparison: CP-690,550 100 mg vs Placebo; 16 hours post-dose; Test type: Superiority; Least Squares Mean Difference = 2.10, 90% CI 2-sided [-0.17 to 4.38]
Statistical Analysis 9: Comparison: CP-690,550 100 mg vs Placebo; 24 hours post-dose; Test type: Superiority; Least Squares Mean Difference = 0.79, 90% CI 2-sided [-1.49 to 3.06]

12. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] for CP-690,550
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: Pharmacokinetic (PK) parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
nanogram*hour/milliliter (ng*hr/mL) | 2682.6 (778.15)

13. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for CP-690,550
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
ng*hr/mL | 2669.7 (771.02)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of CP-690,550
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 13
Measure: Geometric Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
nanogram/milliliter (ng/mL) | 563.5 (199.23)

15. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for CP-690,550
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Groups:
- CP-690,550 100 mg: Single oral dose of CP-690,550 100 mg (5 x 20 mg tablets) in all intervention periods.
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
hours | 1.000 [0.30 to 4.08]

16. Secondary Outcome: Plasma Decay Half-Life (t1/2) of CP-690,550
Description: Plasma decay half-life is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
hours | 3.284 (0.4871)

17. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of CP-690,550 by Cytochrome P450 2C19 (CYP2C19) Genotype
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). Variation in CYP2C19 gene affected the pharmacokinetics of CP-690,550. AUC (0 - ∞) categorized by genotype into poor metabolizer, extensive metabolizer and ultra extensive metabolizer of CYP2C19.
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Here 'number analyzed' signifies those participants who were evaluable in each specific category.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
ng*hr/mL
  Poor Metabolizer: number analyzed (Participants) | 6
  Poor Metabolizer | 3127.5 (373.18)
  Extensive Metabolizer: number analyzed (Participants) | 52
  Extensive Metabolizer | 2683.5 (787.75)
  Ultra Extensive Metabolizer: number analyzed (Participants) | 2
  Ultra Extensive Metabolizer | 1677.7 (637.68)

18. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of CP-690,550 by CYP2C19 Genotype
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). Variation in CYP2C19 gene affected the pharmacokinetics of CP-690,550. AUClast categorized by genotype as poor metabolizer, extensive metabolizer and ultra extensive metabolizer of CYP2C19.
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
ng*hr/mL
  Poor Metabolizer: number analyzed (Participants) | 6
  Poor Metabolizer | 3114.3 (366.68)
  Extensive Metabolizer: number analyzed (Participants) | 52
  Extensive Metabolizer | 2670.2 (780.41)
  Ultra Extensive Metabolizer: number analyzed (Participants) | 2
  Ultra Extensive Metabolizer | 1673.1 (636.30)

19. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of CP-690,550 by CYP2C19 Genotype
Description: Variation in CYP2C19 gene affected the pharmacokinetics of CP-690,550. Cmax categorized by genotype as poor metabolizer, extensive metabolizer and ultra extensive metabolizer of CYP2C19.
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
ng/mL
  Poor Metabolizer: number analyzed (Participants) | 6
  Poor Metabolizer | 647.4 (281.69)
  Extensive Metabolizer: number analyzed (Participants) | 52
  Extensive Metabolizer | 565.0 (185.62)
  Ultra Extensive Metabolizer: number analyzed (Participants) | 2
  Ultra Extensive Metabolizer | 346.9 (214.25)

20. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of CP-690,550 by CYP2C19 Genotype
Description: Variation in CYP2C19 gene affected the pharmacokinetics of CP-690,550. Tmax categorized by genotype as poor metabolizer, extensive metabolizer and ultra extensive metabolizer of CYP2C19.
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
hours
  Poor Metabolizer: number analyzed (Participants) | 6
  Poor Metabolizer | 0.500 [0.30 to 4.03]
  Extensive Metabolizer: number analyzed (Participants) | 52
  Extensive Metabolizer | 1.000 [0.30 to 4.08]
  Ultra Extensive Metabolizer: number analyzed (Participants) | 2
  Ultra Extensive Metabolizer | 2.000 [2.00 to 2.00]

21. Secondary Outcome: Plasma Decay Half-Life (t1/2) of CP-690,550 by CYP2C19 Genotype
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Variation in CYP2C19 gene affected the pharmacokinetics of CP-690,550. t1/2 categorized by genotype as poor metabolizer, extensive metabolizer and ultra extensive metabolizer of CYP2C19.
Time Frame: 0 (pre-dose), and 0.25, 0.5, 1, 2, 4, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CP-690,550 100 mg
Number analyzed (Participants) | 60
hours
  Poor Metabolizer: number analyzed (Participants) | 6
  Poor Metabolizer | 3.005 (0.3566)
  Extensive Metabolizer: number analyzed (Participants) | 52
  Extensive Metabolizer | 3.320 (0.5006)
  Ultra Extensive Metabolizer: number analyzed (Participants) | 2
  Ultra Extensive Metabolizer | 3.201 (0.1821)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant , or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- Moxifloxacin: Single oral dose of moxifloxacin 400 mg tablet in any intervention period.
Arm/Group | CP-690,550 100 mg | Placebo | Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 32/60 | 6/60 | 10/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 100 mg (N=60) | Placebo (N=60) | Moxifloxacin (N=60)
Palpitations (Cardiac disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 17 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2
Headache (Nervous system disorders) | 17 | 1 | 2
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.